CLINICAL TRIAL: NCT05753579
Title: Is Regression Possible in Lumbal Disc Herniation Through Spinal Mobilization Applications? Double-Blind Randomized Controlled Clinical Trial
Brief Title: Is Regression Possible in Lumbal Disc Herniation With Spinal Mobilization Applications?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10879717-050.01.04
Record Dates: First submitted 2023-02-05; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Intervertebral Disc Displacement; Disk Herniated Lumbar; Disc Herniation
Keywords: Lumbar disc herniation; Manual Therapies; Mobilization; Stabilization Exercises
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: This study was designed as a double-blind randomized controlled clinical trial. In order to carry out the prospectively designed study, ethics committee approval was obtained from the Non-Interventional Clinical Research Ethics Committee of Muş Alparslan University with the decision numbered 21 taken at the meeting dated 29.12.2020 and numbered 15. Informed consent was obtained from all patients included in the study before the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible patients were divided into two groups using the closed envelope method at a ratio of 1:1. The patients did not know which group they were in. This grouping was unknown to the radiologist performing the evaluation and the statistician performing the data analysis. Mobilization applications and other clinical tests were performed by the same physiotherapist in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): In our study, stabilization exercises were applied to the patients in the control group. The treatment was applied two days a week for five weeks, for a total of ten sessions. After the end of the treatment, stabilization exercises were recommended as a home exercise program until the follow-up evaluation at the third month. A telephone connection was established with the patients once a week and the home program was followed up.Stabilization exercises: It is an approach that is combined with diaphragmatic breathing and activates the passive. The stabilization exercise program was applied in three phases and was progressed in line with the developments in the patients.
  Interventions: Behavioral: Stabilization Exercise
- Intervention Group (Experimental): In our study, stabilization exercises and spinal mobilization practices were performed to the patients in the intervention group. The treatment was applied two days a week for five weeks, for a total of ten sessions. After the end of the treatment, stabilization exercises were recommended as a home exercise program until the follow-up evaluation at the third month. A telephone connection was established with the patients once a week and the home program was followed up.Mobilization applications were applied at Maitland IV degree as standard.Three mobilization methods were applied Anterior-Posterior Lumbal Spinal Mobilization Lumbal Spinal Rotational Mobilization Joint Mobilization in Lumbal Flexion Position
  Interventions: Behavioral: Spinal Mobilization; Behavioral: Stabilization Exercise

INTERVENTIONS:
Behavioral: Spinal Mobilization — Mobilization applications are passive movements that do not involve pushing or stimuli, applied within the range of motion or up to the physiological range of motion.
  Arms: Intervention Group
Behavioral: Stabilization Exercise — Diyafragmatik solunum ile kombine edilen, pasif-aktif kas iskelet sistemi ve nöral sistemi aktive eden bir yaklaşımdır. Bu yaklaşımda derin çekirdek kaslar olarak transversus abdominis, multifudus kasları aktive edilmektedir

SUMMARY:
Spinal mobilization methods are passive maneuvers that are made lighter and do not exceed the physiological range of motion in order to increase joint mobility. Mobilization applications are easier and safer than manipulation applications involving forceful pushing. Although there are many literatures reporting the therapeutic efficacy of long-term mobilization applications on LDH, there is no study on the effect of applications on radiological findings of LDH.

In the light of the information mentioned above, the aim of this study is; To examine the effect of mobilization applications on radiological findings and functional level in patients with LDH

DETAILED DESCRIPTION:
Disc herniation is the herniation of the nucleus pulposus, which is the disc material, into the spinal canal along the fibers of the annulus fibrosus. Spinal herniations that affect the whole spine are most common in the lumbar region, and most often in the L4-L5 and L5-S1 levels in this region. Lumbar disc herniation (LDH) is a common cause of low back pain, radicular pain, and radiculopathy, resulting in disability. Depending on the size of the herniation, the nerve is compressed in the lateral recess or in the foraminal or extraforaminal space. The pathophysiology of pain includes direct nerve root compression and local inflammation. Scientists have found that myelography is not as sensitive as magnetic resonance imaging (MRI) in diagnosing lumbar disc herniation, and MRI has a higher positivity rate. Compared with computed tomography, it has more imaging parameters, multiple tissue variable functions, more flexible and comprehensive, no radiation and no harm to the human body, and the diagnostic accuracy is better than CT scanning. Because of these advantages, MRI is the gold standard imaging method in the diagnosis of LDH. There are various treatment options available for LDH patients. These are basically divided into 2 categories: surgical and conservative care. Conservative care includes oral medications, corticosteroid and anesthetic infiltrations (nerve root injections), bed rest, exercise therapy, flexion/distraction therapy, manipulation and mobilization.Mobilization applications are passive movements that do not involve pushing or stimuli, applied within the range of motion or up to the physiological range of motion. Mobilization has mechanical effects such as increasing tissue flexibility, separating adhesions, relieving joint limitation and reducing intra-articular pressure. Evidence suggests that mobilizations cause a neurophysiological effect that results in sympathetic arousal, reduced neural mechanical sensitivity, mechanical hypoalgesia, and normalized muscle activity, endurance, and pain-free strength.There are many studies on the clinical use of mobilization methods. While most of these studies examine the effects of mobilization on pain and functional status in patients with low back pain, there are also studies examining the effects of mobilization on pain, functional status and activities of daily living in patients with LDH. In the literature, it has been determined that regression in the lumbar disc herniation distance is achieved with conservative treatment and medical treatment approaches. It is observed that there are studies examining the effect of manipulation on the herniation distance, which is one of the non-invasive Spinal Decompression Therapy method and Manual therapy methods. However, there is no study in the literature investigating the regression of spinal mobilization applications in LDH patients.The aim of our study is to examine the effects of spinal mobilization applications applied in three different planes in addition to stabilization exercises on radiological findings such as herniation distance, disc height and facet joint distance in LDH patients. Apart from radiological findings, it was also aimed to investigate the effects of patients on functional status, pain and flexibility.

ELIGIBILITY:
Inclusion Criteria

* It was determined as being diagnosed with LDH by MR by a physical therapy physician
* Having pain of at least 3 levels or more according to the Visual Analogue Scale
* Being between the ages of 18-65.

Exclusion Criteria

* History of spinal surgery
* History of autoimmune disease (ankylosing spondylitis, rheumatoid arthritis or other)
* Spondylolysis and spondylolisthesis
* Spinal fracture
* Heart pathology
* History of stroke,
* Cauda equina syndrome
* Continuous use of pain medication
* Spinal inflammation,
* Spinal tumor
* Covid
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Radiologic Assessment | The change of the disc height, herniation thickness and ZGAP (facet joint distance) were measured twice by a radiology expert before and after treatment
  MRI examinations were performed before and after treatment in the same center. In both evaluations, the specialist radiologist did not know which group the patient was in. T2 and T1-weighted sagittal sections and T2-weighted axial sections were used as a basis for MRI evaluations. Disc height, hernia thickness and facet joint distance were evaluated in millimeters (mm). In case of herniation at different levels in the same person, the evaluation was performed on the level with the highest herniation degree. All MRI scans were done between 16 and 18 pm during the day.

SECONDARY OUTCOMES:
Functional Assessment | The change of functional capacity of patients participating in the study was assessed before treatment, through treatment completion, an average of 1 week and 3 months after treatment using the Oswestry Low Back Pain Disability Questionnaire.
  Back Performance Scale (BPS): It is a scale used to detect performance that differs depending on low back pain. The scale consists of 5 questions and 4 options valued between 0-3 for each question. The result is obtained by summing the answers given to the questions. The higher the score, the lower the performance.
Pain Assessment | The change of pain assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Visual Analog Scale (VAS): It is used to convert some values that cannot be measured numerically to digital. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.
Range Of Motion Assesment | The change of range of motion assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Straight Leg Raise Test: In the evaluation of straight leg lift, the inclinometer was placed anterior to the tibia while the patient was lying on his back. The inclinometer was reset, the patient was asked to raise his leg and the value displayed on the inclinometer was recorded at the last point.
Flexibility Assessment | The change of flexibility assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Sit and Reach Test: The person being tested was asked to come to a long sitting position with the knees straight and rest the soles of their feet flat on the bottom of the test board. The feet were positioned to be approximately shoulder-width apart, and the patient reached forward from the waist and hips with elbows, wrists and fingers tense. Care was taken to keep the knees straight during the test. The person being tested pushed forward the measuring board on the test bench with his fingers and waited for 1-2 seconds at the end point. The point where the feet made contact with the test bench was taken as the starting point, the 0 point. It was measured from the fingertip to the starting point and recorded in cm as '-' if it is in front of 0 point and '+' if it is behind.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Taşkaya, Principal Investigator — Muş Alparslan University
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No